CLINICAL TRIAL: NCT04062175
Title: Efficacy of Adding Azithromycin to Cephalosporin for the Prophylaxis Against Infectious Morbidity Following Cesarean Delivery in High Risk Women
Brief Title: Efficacy of Adding Azithromycin to Cephalosporin Before Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada fayed hashem el sharkawy, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 55
Record Dates: First submitted 2019-08-13; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Wound Sepsis
MeSH Terms: interventions — Cephalosporins; Azithromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cephalosporin arm (Active Comparator): 72 women will receive single antibiotic chemotheraby first generation cephalosporin (cefazolin) 2 gm iv within 30 minutes before skin incision
  Interventions: Drug: cephalosporin
- cephalosporin +azithromycin arm (Active Comparator): 72 women will receive combined antibiotic chemotherapy azithromycin (Azrolid) 1 gm single oral dose 2 hours before cesarean delivery + cephalosporin(Cefazolin) 2 gm iv within 30 minutes before skin incision
  Interventions: Drug: cephalosporin; Drug: Azithromycin Tablets

INTERVENTIONS:
Drug: cephalosporin — 72 women will receive single antibiotic chemotherapy(Cefazolin) 2 gm iv within 30 minutes before skin incision
Drug: Azithromycin Tablets — 72 women will receive combined antibiotic chemotherapy azithromycin(Azrolid) 1 gm single oral dose 2 hours before cesarean delivery +cephalosporin(Cefazolin) 2 gm iv within 30 minutes before skin incision
  Arms: cephalosporin +azithromycin arm

SUMMARY:
efficacy of adding azithromycin to cephalosporin before cesarean delivery

DETAILED DESCRIPTION:
efficacy of adding azithromycin to cephalosporin for the prophylaxis against infectious morbidity following cesarean delivery in high risk women

ELIGIBILITY:
Inclusion Criteria:

* age between 17 and 39 years
* gestaional age between 37 to 42 weeks
* elective cesarean delivery
* obese women

Exclusion Criteria:

* diabetic women on corticosteroids
* intraopertaive complication in previous section
* history of septic woun
* prelabour rupture of membrane >12 hours

Ages: 17 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
% of women with wound infection | after 14 days post cesarean delivery
  superficial and deep surgical site wound infection will be looked for by laboratory confirmation

SECONDARY OUTCOMES:
% of women with postpartum endometritis | after 14 days post cesarean delivery
  fever, abdominal pain , uterine tenderness will be looked for

CONTACTS AND LOCATIONS:
Overall Officials: Reda Mokhtar, MD, Principal Investigator — AinShams university ,egypt el abbasia
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No